CLINICAL TRIAL: NCT06687876
Title: Metformin as a Metabolic Intervention in Oesophageal Adenocarcinomas to Improve Response to Neoadjuvant Chemoradiotherapy.
Acronym: MEMENTO
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Cancer Center Amsterdam Research Foundation (Unknown)
Responsible Party: Principal Investigator, Sarah Derks, MD PhD, Amsterdam UMC, location VUmc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024.0935; 2024-511626-30-00 (EU CTIS Number)
Record Dates: First submitted 2024-11-05; First posted 2024-11-14 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Oesophageal Adenocarcinoma; Tumor Microenvironment
Keywords: metabolic intervention; adenocarcinoma; oesophageal cancer; metformin; tumor microenvironment; neoadjuvant chemoradiotherapy
MeSH Terms: conditions — Adenocarcinoma Of Esophagus; Adenocarcinoma; Esophageal Neoplasms | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Metformin (Experimental): 1000 mg (twice a day 500 mg) metformin orally will be administered during a 2-week period. This is followed by the standard of care, which is neoadjuvant chemoradiotherapy, involving paclitaxel (50 mg/m2), carboplatin (AUC=2), and radiotherapy (23 x 1.8 Gy over five weeks) followed by surgical resection.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Twice a day 500mg of metfomrin orally (1000mg/day) during a 2-week period.
  Other Names: Glucient

SUMMARY:
The primary objective of this study is to investigate whether two weeks of metformin treatment can activate the tumour microenvironment in patients with stage II and III oesophageal adenocarcinomas.

DETAILED DESCRIPTION:
Worldwide oesophageal adenocarcinoma (OAC) is one of the most deadly cancers. Even in case of non-metastatic disease, when patients are treated with neoadjuvant chemoradiotherapy (nCRT) and a surgical resection, around 50% of patients suffer from recurrent disease which is associated with a poor prognosis. While 23% of OACs have a complete histopathological response after nCRT, 18-35% lack any effect of nCRT. Previously, we have identified that a complete pathological response to nCRT is associated with an active tumour immune microenvironment (TIME) characterized by high intratumoral T cell levels and a higher CD3:CD163 ratio.

To improve response to nCRT we need to identify and target the mechanisms OACs use to suppress the TIME. Using spatial transcriptomics to identify differences between OACs with a T cell-dominant and a T cell-excluded microenvironment, we identified fatty acid oxidation (FAO) as central feature of T cell low OACs (unpublished data). This is an interesting observation as lipid metabolism is strongly associated with an immunosuppressive microenvironment. Metabolic re-programming by drugs such as metformin has shown to be a promising strategy to reactivate the anti-tumour immune response in other cancer types.

Over the past decade, metformin has been associated with a beneficial effect in cancer treatment as it has shown to decrease the risk of various cancer types in diabetic patients. More recent, metformin treatment has shown to increase the number of CD8+ tumour infiltrating lymphocytes by preventing apoptosis of these lymphocytes in cancers such as oesophageal squamous cell carcinomas. In addition, metformin can reduce M2-like macrophage polarization due to changes in cytokine expression in cancer cells and thereby stimulate a more pro-inflammatory TIME. In this study we want to investigate the effect of metformin on the TIME in patients with OACs using pre- and post-treatment tumour biopsies prior to nCRT.

ELIGIBILITY:
Inclusion Criteria:

* Surgical resectable (<T4b, N0 or N+, M0), and histologically proven adenocarcinoma of the oesophagus or gastro-oesophageal junction planning to undergo neoadjuvant chemoradiotherapy.
* Adult patients (age ≥ 18 years).
* ECOG performance status 0 or 1 (cf. Appendix A).
* Adequate hematological, renal and hepatic functions defined as:

  * Absolute Neutrophil Count ≥ 1.5 x 10^9/L
  * Platelets ≥ 100 x 10^9/L
  * Hemoglobin ≥ 5.6 mmol
  * Total bilirubin ≤ 1.5 x upper normal limit
  * Creatinine clearance (Cockroft) > 30 ml/min
* Patients must be willing to undergo two endoscopies for investigational purposes.
* Written, voluntary informed consent.
* Patients must be accessible to follow up and management in the treatment center.

Exclusion Criteria:

* Patients diagnosed with diabetes mellitus type 1 or 2 receiving anti-diabetic drugs.
* Patients prescribed metformin or another anti-diabetic drug for any reason.
* Patients allergic or intolerant to metformin.
* Excessive alcohol consumption.
* Use of OCT1/OCT2 inhibitors (e.g. verapamil, cimetidine, dolutegravir, isavuonazol, trimethoprim, vandetanib, crizotinib and Olaparib).
* Use of OCT1/OCT2 inducers (e.g. rifampicine).
* Use of immunosuppressive medication (corticosteroids, cyclosporine, tacrolimus, sirolimus, everolimus, cyclophosphamide).
* Previous systemic therapy or radiotherapy on the oesophagus.
* Severe renal impairment (CLcr ≤ 30 ml/min).
* Past (within 5 years) or current history of malignancy other than entry diagnosis interfering with prognosis of oesophageal cancer.
* Previous systemic therapy for other forms of cancer within the last six months.
* Patients with prior allogeneic stem cell or solid organ transplantation
* Pregnancy (positive serum pregnancy test), planning to become pregnant, and lactation.
* Clinically significant cardiovascular disease (including myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia) precluding major surgery.
* Pulmonary fibrosis, active, non-infectious pneumonitis and/or severely impaired lung function precluding major surgery and/or radiation.
* Serious underlying medical condition which would impair the ability of the patient to receive the planned treatment, including prior allergic reactions to drugs containing Cremophor, such as teniposide or cyclosporine.
* Dementia or altered mental status that would prohibit the understanding and giving of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2025-03-09 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
activation of the tumour immune microenvironment after two week metformin treatment. | at enrollment and at end of metformin treatment at 2 weeks.
  Activation of the tumor immune microenvironment measured by M2 to M1 polarization, CD8 intratumoral T cell infiltration and an increase of CD3 to CD163 ratio when comparing tumor biopsies from before and after treatment.

SECONDARY OUTCOMES:
Tolerability and toxicity of metformin | From starting treatment to end of treatment at 7 weeks.
  Adverse events based on Common Toxicity Criteria for Adverse Events
Metabolic change of cancer cells with SCENITH analysis. | at enrollment and at end of metformin treatment at 2 weeks
  To determine whether SCENITH can be used to assay the change in metabolic state.
Pathological response | After surgery, approximately 16 weeks after enrollment.
  According to the Mandard criteria.
Progression-free survival (PFS). | 60 months
  Assess the PFS of patients within the study
Overall survival (OS) | 60 months
  Determine overall survival of patients within the study

OTHER OUTCOMES:
Can metformin induce a metabolic switch in macrophages, T cells and cancer cells. | 20 months
  Using single cell RNA sequencing or SCENITH analysis.
Change in subgroups in peripheral blood mononuclear cells (PMBCs) after metformin treatment. | 20 months
  Are the changes to the tumour immune microenvironment also detected in subgroups of peripheral blood mononuclear cells (PBMCs) taken at the same time points.
Establish immune cell co-cultures with primary tumour cells and investigate the cell interactions and anti-tumour responses in presence of metformin. | 20 months
  Establish autologous immune cell co-cultures with primary tumor cells to investigate immune cell-tumor cell interactions and anti-tumour responses in the presence of metformin.
Cytokine release profile measured in serum before and after metformin treatment. | 20 months
  Determine changes in cytokine expression in serum before and after metformin treatment.
changes in ctDNA in patient plasma before and after metformin treatment. | 20 months
  To evaluate changes in the presence of circulating tumour DNA (ctDNA) extracted from patient plasma and their correlation with pathological response and survival.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Derks, MD PhD, Principal Investigator — Amsterdam UMC, location VUmc; Hanneke W.M. van Laarhoven, MD, PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- Amsterdam UMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
It is undecided.